CLINICAL TRIAL: NCT03937843
Title: Reduced Intensity Radio-chemotherapy for Stage IIA/B Seminoma. A Multicenter, Open Label Phase II Trial With Two Cohorts
Brief Title: Reduced Intensity Radio-chemotherapy for Stage IIA/B Seminoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Collaborators: German Testicular Cancer Study Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAKK 01/18; 2019-000514-11 (EudraCT Number)
Record Dates: First submitted 2019-04-29; First posted 2019-05-06 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Seminoma; Testicular Cancer
Keywords: Seminoma; Stage IIA/B seminoma; Radio-chemotherapy; Phase II trial; Testicular Cancer
MeSH Terms: conditions — Seminoma; Testicular Neoplasms | interventions — Carboplatin; Cisplatin; Etoposide

STUDY DESIGN:
Intervention Model Description: A multicenter, open label phase II trial with two cohorts
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm with 2 cohorts (Experimental): Cohort 1: Primary stage IIA and recurrent stage IIA seminoma after active surveillance for stage I:
  * Within 7 days after registration, the patients will receive one infusion of carboplatin AUC (Area under the curve) 7 at day 1 of trial treatment, followed 3 weeks later by 12 x 2 Gy involved-node radiation therapy (RT). RT should ideally start on day 22 (range: day 19-25) from the date of carboplatin administration, preferably on a Monday.
  Cohort 2: Primary stage IIB and recurrent stage IIB seminoma after active surveillance for stage I OR stage IIA/B seminoma after adjuvant carboplatin or radiotherapy for stage I:
  * Within 7 days after registration, the patients will receive one cycle of etoposide 100 mg/m2/d + cisplatin 20 mg/m2/d at days 1 to 5 of trial treatment, followed 3 weeks later by 15 x 2 Gy involved-node radiation therapy. RT should ideally start on day 22 (range: day 19-25) from the date of chemotherapy start, preferably on a Monday.
  Interventions: Drug: Carboplatin; Drug: Cisplatin; Drug: Etoposide

INTERVENTIONS:
Drug: Carboplatin — Patients in cohort 1 will receive a 60-minute i.v. infusion of carboplatin AUC 7 at day 1 of treatment.
Drug: Cisplatin — Patients in cohort 2 will receive on day 1 to day 5:
  * a 60-minutes i.v. infusion of etoposide 100mg/m2 per day followed by
  * a 60-120 minutes i.v. infusion of cisplatin 20mg/m2 per day.
Drug: Etoposide — Patients in cohort 2 will receive on day 1 to day 5:
  * a 60-minutes i.v. infusion of etoposide 100mg/m2 per day followed by
  * a 60-120 minutes i.v. infusion of cisplatin 20mg/m2 per day.

SUMMARY:
The trial investigates a stage-adapted (stage IIA or IIB) de-escalation of the standard treatments in the context of a multimodality treatment with chemo- and radiotherapy in seminoma patients. The goal is to safely de-escalate treatment while maintaining/enhancing efficacy, which is not a standard practice yet.

DETAILED DESCRIPTION:
Therapy de-escalation in stage IIA/B seminoma represents an unmet need in clinical practice; efficacy of modern standard of care therapies for these patients is high and only a few patients show disease recurrence but short- and long-term toxicities are a major concern. The magnitude of long-term toxicities is often associated with the intensity of the prescribed treatment modality. A higher cumulative dose of chemotherapy agents and radiation dose has been linked to a sharp increase in long-term sequelae. Combining treatment modalities and diversifying toxicity may thus provide an opportunity to limit long-term treatment sequelae.

In this trial carboplatin, cisplatin and etoposide are the Investigational Medicine Products (IMPs). They are all medications with a marketing authorization for several solid tumor types and are standard practice in the treatment of testicular cancer in Switzerland and in the European Union (EU).

Radiotherapy is also a standard therapy in this indication.

However, the trial investigates a stage-adapted (stage IIA or IIB) de-escalation of these standard treatments in the context of a multimodality treatment with chemo- and radiotherapy. The goal is to safely de-escalate treatment while maintaining/enhancing efficacy, which is not a standard practice yet.

The SAKK 01/18 trial is designed with the aim to answer these three questions:

* Can the dose of involved-node radiotherapy be safely reduced in the context of multimodality treatment with chemo- and radiotherapy?
* Can a more potent chemotherapy in the form of cisplatin/etoposide reduce the rate of distant failure in comparison to carboplatin?
* Can a combination of cisplatin/etoposide and involved-node radiotherapy pose a potent treatment regime for patients with recurrence after adjuvant carboplatin or radiotherapy for stage I seminoma? Furthermore, as active surveillance is becoming standard of care in stage I seminoma, it is projected that the amount of patients in need of treatment with stage IIA/B disease will rise, due to more patients developing disease progression during active surveillance.

The trial design, trial treatment and trial specifics are a consensus among the Swiss Urogenital Tumors Project Group and the Swiss Radio-oncology Section from the Swiss Group for Clinical Cancer Research (SAKK) and the German Testicular Cancer Study Group (GTCSG).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent according to ICH/GCP (International Council on Harmonization/Good Clinical Practice) regulations before registration and prior to any trial specific procedures
* Histologically confirmed classical seminoma treated with primary inguinal orchidectomy or partial orchidectomy
* Patients with a seminoma stage IIA or IIB, either newly diagnosed or recurrent after primary active surveillance, adjuvant carboplatin or radiotherapy for stage I disease. The tumor stage is pT1-4 cN1-2 cM0 according to UICC TNM 8th edition 2016. Patients with a recurrent seminoma stage IIA or IIB are only eligible in case of progression under active surveillance or recurrence after adjuvant carboplatin or radiotherapy for stage I disease
* Stage IIA, in patients with equivocal lymph node enlargement, needs to be confirmed with a repeated CT/MRI scan of the abdomen (suggested timeframe: 4 weeks after the previous scan) in order to rule out false positive lymph node enlargement.

Patients with a prior malignancy treated with curative intention are eligible if all treatment of that malignancy was completed at least 5 years before registration and the patient has no evidence of disease at registration. Less than 5 years is acceptable for malignancies with low risk of recurrence and/or no late recurrence. Patients with a germ cell neoplasia in situ (GCNIS) or contralateral localized treated seminoma are eligible

* Diagnostic CT or MRI or FDG-PET-CT of the chest, abdomen and pelvis within 28 days prior to registration, showing stage IIA/B disease. I.v. contrast medium has to be administered
* Age ≥ 18 years
* WHO performance status 0-2
* Baseline PRO questionnaires have been completed
* Adequate bone marrow function: neutrophil count ≥ 1.0 x 109/L, platelet count ≥ 100x 109/L
* Adequate renal function: creatinine clearance ≥ 60 ml/min calculated according to the CKD-EPI (Chronic Kidney Disease Epidemiology Collaboration) formula
* Patient agrees to use highly effective contraception and not to donate sperm or to father a child during trial treatment and during 12 months thereafter. Patient has been proposed sperm conservation.

Exclusion criteria

* Any other histological component than seminoma
* Elevated levels of Alpha-1-Fetoprotein AFP (≥ 2x ULN)
* Involved nodes (metastatic) in previously irradiated localizations in the abdomen or pelvis
* Any anti-cancer therapy after primary tumor resection in patients presenting with primary stage IIA/B seminoma
* Any serious underlying medical condition (i.e. current renal insufficiency, severe hepatic insufficiency, severe bone marrow dysfunction, tumor bleeding, major hearing defects) or serious co-morbidity which could impair the ability of the patient to participate in the trial (according to investigator's judgment)
* Any treatment in a clinical trial within 28 days prior to registration
* Any concomitant drugs contraindicated for use with the trial drugs according to the approved product information or contraindicated for use with radiotherapy
* Known hypersensitivity to trial drugs or to any component of the trial drugs
* Any other serious underlying medical, psychiatric, psychological, familial or geographical condition, which in the judgment of the investigator may interfere with the planned staging, treatment and follow-up, affect patient compliance or place the patient at high risk from treatment-related complications.

Additional German specific exclusion criteria - not to be considered for Swiss patients

* Patient who is dependent on the sponsor or the investigators according to ICH/GCP E6(R2), guideline
* Patient who has been committed to an institution by virtue of an order issued either by the judicial or the administrative authorities according to § 40a (2) AMG.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2019-07-29 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2046-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) at 3 years | From the date of registration until the date of progressive disease, relapse or death, whichever occurs first, assessed up to 3 years after registration
  PFS is defined as the time from registration until one of the following events occurs:
  * Progressive disease or relapse, defined as progression according to the modified trial-specific version of RECIST 1.1 or a rising level of the tumor marker beta-hCG (beta human chorionic gonadotropin) over the ULN (Upper limit of normal), confirmed by a second measurement. Presence of non-seminoma germ cell tumor has to be excluded in the latter case
  * Death from any cause.

SECONDARY OUTCOMES:
Response rate (RR) | at 3 months and 3 years after registration
  The response is categorized according to the modified trial-specific version of RECIST 1.1 measurability criteria as: complete remission (CR), partial remission (PR), stable disease (SD), progressive disease (PD).
  The response rate is defined as proportion of patients with CR or PR on imaging assessment and without rising beta-hCG. Patients with CR, PR and SD on imaging assessment, but with confirmed rising beta-hCG will not be counted as responders, if the presence on non-seminoma germ cell tumor was excluded. Response rate will be evaluated at 3 months and 3 years after registration.
Progression free survival (PFS) | From the date of registration until the date of progressive disease, relapse or death, whichever occurs first, assessed up to 20 years after registration
Time to progression (TTP) | From the date of registration until the date of progressive disease, relapse or death due to progression, whichever occurs first, assessed up to 20 years after registration
  TTP is defined as the time from registration until documented PD or relapse according to the modified trial-specific version of RECIST 1.1 or death due to progression, whichever occurs first.
  Patients without an event at the time of analysis and patients starting a new anticancer therapy in the absence of an event will be censored at the date of the last tumor assessment showing non-progression before the start of a new therapy, if any.
Overall Survival (OS) | From the date of registration until the date of death from any cause, assessed up to 20 years after registration
  OS is defined as the time from registration to the date of death from any cause. Patients who did not experience an event will be censored at the last known time they were known to be alive.
Seminoma-specific survival | From the date of registration until the date of death due to seminoma, assessed up to 20 years after registration
  Seminoma-specific survival is defined as the time from registration to the date of death due to seminoma. Patients who did not experience an event will be censored at the last known time they were known to be alive.
Time to distant metastasis | From the date of registration until the date of first occurrence of distant metastasis, assessed up to 20 years after registration
  Time to distant metastasis is defined as the time from registration until first occurrence of distant metastasis. Patients not experiencing an event will be censored at the date of the last available assessment.
Time to next treatment | From the date of registration until the date of start of any new anticancer therapy for progressive seminoma, assessed up to 20 years after registration
  Time to next treatment is defined as the time from registration to the start of any new anticancer therapy for progressive seminoma. Patients not receiving any new treatment are censored at the last date they were known to be alive.
Localization of progression | at the date of the first occurrence of progressive disease, assessed from registration up to 20 years after registration
  The localization of progression is defined as the first localization where progressive disease is detected. It is divided into the following sites:
  * Initially involved lymph node area
  * Non-initially involved paraaortic & pelvic lymph node area
  * Supradiaphragmatic lymph node area
  * Organ involvement (lung, liver, bones, etc.)
  * Multiple sites simultaneously
Method of detection of progression | at the date of the first occurrence of progressive disease, assessed from registration up to 20 years after registration
  The method of detection of progression is defined as the first method used to detect the first progression event and comprises the following categories:
  * Physical examination (inspection, palpation, etc.)
  * Rising beta-hCG tumor marker
  * CT imaging
  * Ultrasound imaging
  * X-ray imaging
  * Other imaging (e. g. MRI, PET-CT)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandros Papachristofilou, MD, Study Chair — Universitätsspital Basel
Locations (19):
- Germany (9):
  - Rotkreuzklinikum München, München, München
  - Vivantes Klinikum Am Urban, Berlin
  - Helios Klinikum Berlin-Buch, Berlin
  - Evang. Kliniken Essen-Mitte, Essen
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - ASKLEPIOS Kliniken, Hamburg
  - RKH Klinikum Ludwigsburg, Ludwigsburg
  - Universitätsklinikum Tübingen, Tübingen
  - Universitätsklinikum Ulm, Ulm
- Switzerland (10):
  - Universitaetsspital-Basel, Basel
  - Istituto Oncologico della Svizzera Italiana (IOSI), Bellinzona
  - Inselspital Bern, Bern
  - Kantonsspital Graubuenden, Chur
  - Kantonsspital Graubünden, Chur
  - Centre Hospitalier Universitaire Vaudois CHUV, Lausanne
  - Kantonsspital - St. Gallen, Sankt Gallen
  - Hopital de Sion, Sion
  - Kantonsspital Winterthur, Winterthur
  - UniversitätsSpital Zürich, Zurich